CLINICAL TRIAL: NCT00708136
Title: Effect of Water-Exercise on Balance Function of Healthy Elderly Individuals - A Randomized Control Study
Brief Title: Effect of Water-Exercise on Balance Function of Healthy Elderly Individuals
Acronym: EWEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: itshak Melzer, Ben-gurion Univesity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sor404605ctil; ISRCTN4046
Record Dates: First submitted 2008-06-29; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2005-11

CONDITIONS: Stability; Balance
Keywords: Falls; elderly; Balance; speed of stepping; Stability; ELDERLY FALLERS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: water based training program to improve balance

SUMMARY:
The proposed project is a Randomized Controlled study design. Seniors (age >65) willing to participate in the study will be shortly interviewed to assess eligibility according to the inclusion-exclusion criteria. The first 60 subjects who upon questioning were judged to meet the following inclusion criteria:

1. able to stand independently 90 seconds
2. able to walk 10 meters (with cane if necessary)
3. able to understand verbal instructions.

The exclusion criteria will be:

1. Serious visual impairment
2. Inability to ambulate independently (cane acceptable, walker not).
3. Severely impaired cognitive status (score less then 24 in Mini Mental State Examination).
4. Persons with impaired communication capabilities.

The whole project will be conducted over a period of 24 months. The proposed study is a randomized experimental intervention/ control group design. A total of 60 elderly volunteer subjects will be randomly assigned to two groups, exercise group (30) and control group (30). Twelve training periods will be performed with 8 subjects participating in training during each period (4 exercise groups). The exercise group will meet on 24 occasions over a period of 12 weeks (2 times/week).

Gait and balance function will be tested in both groups with well established measuring techniques before and after the training period. The measuring techniques

1. Medical background variables.
2. Berg Balance Scale.
3. Late life Function and Disability Instrument.
4. Get up and go test - stand up and walk 3 meters turn around and walk back to the chair.
5. Fall Efficacy Scale
6. Fall incidence and fall severity.
7. 6-minute walk test. The control group will not perform any specific balance training during the 12 week period.

These individuals from control will participate in a separate exercise program after the training period.

The water training intervention is performed on different levels where each level reflects different increasing demands on the postural control system. The water exercises also include perturbation exercises that trigger specific reflex-like balance responses. On each level the instructor can instantly modify an exercise to be more or less challenging for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. able to stand independently 90 seconds;
2. able to walk 10 meters (with cane if necessary);
3. able to understand verbal instructions.

Exclusion Criteria:

1. Serious visual impairment;
2. Inability to ambulate independently (cane acceptable, walker not).
3. Severely impaired cognitive status (score less then 24 in Mini Mental State Examination).
4. Persons with impaired communication capabilities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | before and 3 months after Training
Late life Function and Disability Instrument | before and after the training
Get up and go test | before and after 3 month of training
Step execution test under single and dual task | before and 3 months after Training
Stability tests | before and 3 months after Training

CONTACTS AND LOCATIONS:
Overall Officials: Itshak Melzer, PhD, Principal Investigator — Ben-gurion University of the Negev, Beer-Sheva, Israel; dagan Shvartz, MD, Study Chair — Ben-Gurion University of the Negev
Locations (1):
- SorokaUMC, Beersheba, Israel

REFERENCES:
- [Derived] Melzer I, Elbar O, Tsedek I, Oddsson LIe. A water-based training program that include perturbation exercises to improve stepping responses in older adults: study protocol for a randomized controlled cross-over trial. BMC Geriatr. 2008 Aug 17;8:19. doi: 10.1186/1471-2318-8-19. PMID 18706103